CLINICAL TRIAL: NCT05974878
Title: The Effect of the Physiotherapy Program Developed for the Upper Extremity in Diabetic Individuals on Dexterity, Proprioception, and Functionality
Brief Title: The Effect of the Physiotherapy Program for Diabetic Individuals on Dexterity, Proprioception, and Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Zeynep Irem BULUT, Research Assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/45
Record Dates: First submitted 2023-05-18; First posted 2023-08-03 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes; upper extremity; hand; exercise; proprioception; dexterity; functionality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants in this group are going to be in physiotherapy program, which is created specific to diabetic patients, contains;
  * Exercises for stability, flexibility and strength,
  * Exercises which improves wrist proprioception,
  * Exercises for sensation recovery,
  * Mirror therapy and motor imagination
  * Physiotherapy program will be changed in every 3 weeks. Participant will be informed about their disease, about process of healing and will check by phone calls 2 times a week. They will be given recommendations about disease management. Home exercises will be given to this group and will be added new exercises every 3 weeks while physiotherapy program continues.
  Interventions: Other: Exercise
- Control Group (Experimental): Control group will take conventional physiotherapy as in the literature. Diabetic individuals in routine takes aerobic exercise recommendation and resistive exercises. In our study control group will continue 12 sessions of resistive exercise program focused on upper extremity, also aerobic exercise recommendation.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Exercise — * Joints targeted by exercise; bilateral wrist, metacarpophalangeal, proximal and distal interphalangeal joints, elbow and shoulder joints.
  * The muscles targeted by the exercises; lumbricals, iinterosseals, thenar and hypothenar muscles, forearm flexors, forearm extensors, forearm supinators and pronators, elbow flexors and extensors, and shoulder girdle muscles.
  * Content of the exercises; There will be warm-up exercises, pinch grip, full grip, nerve and tendon gliding exercises, exercises that improve proprioception, functional exercises, strengthening exercises and stretching exercises.
  Arms: Treatment Group
Other: Conventional Physiotherapy — For control group there will be aerobic exercise recommendation and resistive exercises focused on upper extremity.
  Arms: Control Group

SUMMARY:
The goal of our research titled "The effect of the exercise program developed for the upper extremity in diabetic individuals on dexterity, grip strength and proprioception" is to examine the effect of the exercise program created for upper extremity problems in diabetic individuals on dexterity, wrist proprioception and upper extremity functionality. Secondary aims of our study; the exercise program created for upper extremity problems; to investigate the effects of grip strength, neuropathic pain, light touch, proprioception, muscle viscoelastic properties, anxiety and depression levels and quality of life of individuals.

The strength of different grip types will be measured, and an evaluation will be made in a short time from the muscle surface with a device called MyotonPro to determine the characteristics of the muscles in hands and arms. In addition to these, 6 separate questionnaires will evaluate the functionality of hands, wrists and upper extremities, pain level, satisfaction level, difficulty level in daily living activities, neuropathic pain problems, depression and anxiety levels and quality of life. In addition, different senses in the upper extremity and hand-wrist will be tested. These measurements will take 1 hour in total and will be repeated 3 times at 6-week intervals. Participant will divide on 2 groups and treatment group will perform exercises with physiotherapist and control group will take conventional physiotherapy program for diabetes. Comparison will be between groups.

DETAILED DESCRIPTION:
* 12 weeks/ 3 days a week/ 40 minutes of physiotherapy program will be planned. Patients will complete the exercises with a physiotherapist once a week, and home programs given as homework according to weekly targets will be checked by phone calls twice a week. In the first session, information about diabetes will be given and training will be given.
* Content of the exercises; There will be warm-up exercises, pinch grip, full grip, nerve and tendon gliding exercises, exercises that improve proprioception, functional exercises, strengthening exercises and stretching exercises. Control group will be in conventional physiotherapy program once a week as treatment group. The program is going to include aerobic exercise recommendation and basic stretching and strengthening exercises focusing upper extremity muscles.

This research will shed light on the rehabilitation programs to be planned for problems involving the hand in individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being diagnosed with Type 2 diabetes according to the criteria of the American Diabetes Association (ADA)

Exclusion Criteria:

* Insufficient cognitive level
* Traumatic nerve injury
* Presence of congenital anomaly in the upper extremity
* Presence of systematic disease (eg rheumatologic)
* Having a problem involving the neurological system
* Having undergone surgery involving the upper extremity in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Proprioception | From enrollment to the end of treatment at 12 weeks, and at 6th week
  35 degrees wrist flexion and 45 degrees wrist extension will be taught to the patient, and the patient will be asked to bring the wrist to the same position with eyes closed, and the angle of deviation will be measured with a goniometer and recorded.
Dexterity | From enrollment to the end of treatment at 12 weeks, and at 6th week
  The 9-Hole Peg Test, which is a valid and reliable assessment method, will be used to evaluate the hand and finger dexterity of the patients. Randomly placing 9 wooden pins on the 9-hole wooden block as quickly as possible and then removing the pins one by one from the wooden block and placing them in the storage section will be recorded by measuring with a stopwatch. By calculating the total time, 20 seconds or more will be considered as a loss of skill.
Functionality | From enrollment to the end of treatment at 12 weeks, and at 6th week
  The Quick Diasbilities of Arm, Shoulder and Hand (DASH) questionnaire will be used to determine the level and symptoms of physical disability in the upper extremity. Higher scores indicate higher disability in the upper extremity. The Michigan Hand Outcome Questionnaire is used to evaluate complaints in the hands of patients. It can evaluate each hand separately and was developed to evaluate the symptoms of all hand disorders. The parameters it evaluates respectively; function, daily activities, work performance, pain, aesthetics, satisfaction. A high score in the pain domain indicates worsening, and a high score in all other domains indicates a better condition. The total score is obtained by summing the results of the affected extremity or, if bilateral extremities are affected, by adding the mean scores of the areas and dividing by six. This questionnaire is valid and reliable for Turkish society.

SECONDARY OUTCOMES:
Grip strength | From enrollment to at the end of treatment at 12 weeks, and at the 6th week
  Grip strength will be evaluated using the Jamar Dynamometer. The average of three attempts for each hand will be recorded in kilograms. This test is a reliable and valid test to evaluate manual grip strength.
Pinch strength | From enrollment to at the end of treatment at 12 weeks, and at the 6th week
  Grip strength will be evaluated using the Jamar Pinchmeter. The average of three attempts for each hand will be recorded in kilograms. This test is a reliable and valid test to evaluate manual grip strength.
Neuropathic pain | From enrollment to at the end of treatment at 12 weeks, and at the 6th week
  Mc Gill Pain Scale Short Form will be used in pain assessment. The scale consists of 3 sub-sections that evaluate the sensory and perceptual aspects of pain, the severity of pain, and whether there is currently pain. In the first part, there are 15 expressions describing pain and it is graded between 0 (absent) and 3 (severe). In the second part, the patient is expected to mark the severity of pain on a linear scale. In the third part, it evaluates whether the patient currently has pain, and if there is pain, its severity is evaluated with a visual comparison scale. The nature of neuropathic pain will be evaluated with the Neuropathic Pain Questionnaire Short Form (NPQ-SF). The NPQ-SF is a tool used to determine whether there is a complaint of neuropathic pain. It has 3 sub-parameters; tingling pain, increased pain and numbness from constant touch.
Sensations | From enrollment to at the end of treatment at 12 weeks, and at the 6th week
  Two-point discrimination and light touch will be evaluated.
  * Two-point separation; will be done using the discriminator. Two-point discrimination is made to determine the shortest distance that can be felt between two separate points on the skin. It is used to measure the fine work ability and sensitivity of the hand.
  * Light touch; It will be evaluated with the Semmes-Weinstein Monofilament Test. The Semmes-Weinstein Monofilament kit consists of 20 nylon monofilament probes. It is a diagnostic test that objectively measures the touch threshold and is used to reveal the sensory level.
Hand muscles viscoelastic properties | From enrollment to at the end of treatment at 12 weeks, and at the 6th week
  Myoton PRO device will be used to evaluate the viscoelastic properties of the muscle. Three measurements will be made by marking the muscles determined from the thenar (Abductor pollicis brevis) and hypothenar region (Abductor digiti minimi). Myoton PRO (Myoton AS, Tallinn, Estonia) is a handheld device that generates a mechanical impulse on the skin above the target structure. The measurement method implemented by Myoton PRO involves a mechanical pulse oscillating under a constant pressure. The oscillation of the tissue under the probe allows the viscoelastic properties of the tissue to be calculated.
Depression level | From enrollment to at the end of treatment at 12 weeks, and at the 6th week
  Beck Depression Scale will be used to determine the level of depression. It was developed by Beck et al., and its validity and reliability study in our country was performed by Hisli. It contains a total of 21 self-evaluation sentences and is measured with a four-point Likert scale. Each item gets progressively increasing points between 0-3 and the total score varies between 0-63. The high total score indicates the high level of depression or its severity. In the Turkish validity and reliability study of the scale, the cut-off point was determined as 17. A study of the cut-off and psychometric properties of the Beck Depression Scale in the adult Turkish population Kapçı et al. made by. A total score of 0-10 = no depression, 11-17 = mild depression, 18-23 = moderate depression, 24 and above = severe depression.
Anxiety level | From enrollment to at the end of treatment at 12 weeks, and at the 6th week
  Beck Anxiety Scale will be used to determine the level of anxiety. This scale is a Likert-type self-assessment scale consisting of 21 items and scored between 0-3. The high total score indicates the high level of anxiety experienced by the person. It was developed by Beck et al., and its validity and reliability study in our country was performed by Ulusoy et al.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep I BULUT, Mac, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Sahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided